CLINICAL TRIAL: NCT04531969
Title: Comparison of Outpatient and Inpatient Spa Therapy in Knee Osteoarthritis
Brief Title: Comparison of Outpatient and Inpatient Spa Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical Med-2
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Spa therapy; Electrotherapy; Ultrasound; Hotpack
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Patients will be aware of group distribution due to the nature of the study. Therefore, the only outcome assessor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient group (Active Comparator): Spa therapy,HP application, deep heater application, and TENS.
  Interventions: Other: Spa therapy and conventional physical therapy
- Outpatient group (Active Comparator): Spa therapy,HP application, deep heater application, and TENS.
  Interventions: Other: Spa therapy and conventional physical therapy

INTERVENTIONS:
Other: Spa therapy and conventional physical therapy — HP application +deep heater application + TENS. HP application: A hotpack wrapped in a towel for 20 minutes will be placed on the knee and surrounding soft tissues.
  Deep heater application: The application will be performed with a therapeutic ultrasound device at a dose of 1.5watt / cm2 for each string for 6 minutes.
  TENS application:TENS device with two electrodes surrounding tendon will be performed for 30 minutes at low-frequency current application.
  Spa therapy: A conventional water bath water at 38 ° C will be applied in the pool for 20 minutes a day.

SUMMARY:
In this study, we aimed to compare the effectiveness of inpatient and outpatient physical therapy modalities and spa combination treatments on pain and functional status in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) has an important place in musculoskeletal diseases and is the most common rheumatic joint disorder characterized by progressive cartilage degeneration. Osteoarthritis of the knee is the most common symptomatic osteoarthritis characterized by chronic knee pain, joint stiffness, limited daily activities, and decreased quality of life.

In this study, it was aimed to compare the effects of inpatient and outpatient applications of HP, US, TENS, spa combination treatments on pain and functional status in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary knee osteoarthritis

Exclusion Criteria:

* Patients who have secondary knee osteoarthritis due to various diseases
* Patients with pronounced pathology in the waist, hip and ankle joint, patients with active tumors
* Patients with febrile infectious disease
* Having had serious surgical operations in the last 6 months
* Patients who have undergone and/or have been injected with intraarticular steroid and hyaluronic acid into the knee joint
* Patients who have received balneotherapy and peloidotherapy in the last one year
* Patients with decompensated organ failure, those with inflammatory disease, those with pregnancy and breastfeeding
* People with neurological diseases such as epilepsy, inner ear hearing aids, pacemakers and other individuals with a small metallic implant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster University (WOMAC) osteoarthritis index | two weeks
  The form consists of three parts (pain, stiffness, and physical function) and 24 questions. High WOMAC values indicate an increase in pain and stiffness and impairment of physical function.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | two weeks
  The patient was asked to mark the severity of his or her pain with active motion on a horizontal line 100 millimeters in length. The intensity of the pain was calculated by measuring the area in which the individual marked between 0 (no pain) and 10 (the most severe pain I felt in my life).
Timed Up and Go (TUG) | two weeks
  The patient starts in a seated position and stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No